CLINICAL TRIAL: NCT03211585
Title: EVALUATION OF THE EFFECT OF THE PERFECTA V-BEAM LASER ON ROSACEA (FACIAL REDNESS, TELANGIECTASIAS AND PHOTODAMAGE)
Brief Title: EVALUATION OF THE EFFECT OF THE PERFECTA V-BEAM LASER ON ROSACEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Device: Perfecta V-Beam laser — This s a single study and a prototype of the FDA-cleared, flashlamp-pumped pulsed-dye laser, that is currently on the market, that has evolved over almost 25 years of continuous development. The broad-spectrum flashlamp pumps energy into a cavity containing liquid dye. The dye is excited resulting in the emission of 595 nm orange light.

SUMMARY:
The purpose of this study is to further quantify the safety and effectiveness of the Syneron-Candela long pulse-duration, extended sub-pulse, larger spot-size prototype Perfecta V-Beam, 595nm laser system for the treatment of facial redness associated with flushing and blushing, or rosacea. The Perfecta laser system is expected to provide effective treatment of rosacea with less bruising or purpura and greater effectiveness than previous generation systems. This study should enable optimization of treatment parameters for using the Perfecta 595nm laser for treating rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a Fitzpatrick skin type of I-IV and have Rosacea as evaluated by the treating physician.
* Subjects must have visible telangiectasia on the side of the face.
* Subjects must be willing and able to comply with all follow-up requirements.
* Subjects must be willing and able to apply sunblock SPF of 30 while exposed to the sun.
* Subject willing to have photographs taken and used in presentations or publications.

Exclusion Criteria:

* Subjects must not have had a previous laser treatment, deep chemical peel in the intended treatment site(s) within 6 months prior to treatment, oral retinoids within 6 months of their inclusion into this study or have ever taken gold therapy.
* Subjects must not have a history of keloid formation.
* Subjects with Fitzpatrick Classification of V or VI (to reduce the risk of hyper-pigmentation).
* Subjects must be willing and able to comply with all follow-up requirements.
* Subjects cannot have vitiligo, a condition where pigment is lost in the skin and white patches appear).
* Subjects not willing to avoid sun exposure or not will to apply sunblock SPF of 30 while exposed to the sun.
* Subject not willing to have photographs taken and used in presentations, publications and marketing material

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The percentage reduction in the facial redness and telangiectasias of rosacea | two months following the final treatment
  The percentage reduction in the facial redness and telangiectasias of rosacea will be determined by the investigators using polarized photography for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bernstein, MD, Principal Investigator — Main Line Center for Laser Surgery